CLINICAL TRIAL: NCT03738813
Title: Feasibility and Efficacy of the Upper Limb Treatment With "Gloreha Aria" in the Hemiplegic Patients: a Randomized Pilot Study
Brief Title: Upper Limb Treatment With "Gloreha Aria" in the Hemiplegic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICS Maugeri - CE 2208
Record Dates: First submitted 2018-08-23; First posted 2018-11-13 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Hemiplegia and/or Hemiparesis Following Stroke; Upper Extremity Injury
MeSH Terms: conditions — Arm Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): The specific hand intervention consisted of 30 sessions, lasting 60 min/ day, for 6 days/week. All patients will be educated by physiotherapist to perform the movements for wrist, hand and arm in complete autonomy.
  In Treatment Group, the movements will be performed using Gloreha ARIA. Gloreha Aria is a sensor-based therapy device designed for motor recovery of impaired upper limb. Gloreha Aria is equipped with sensors that can detect any movements in space: the software processes and displays them on the screen.
  Interventions: Device: Gloreha Aria
- Participants Usual Care (PUC) (Active Comparator): The specific hand intervention consisted of 30 sessions, lasting 60 min/ day, for 6 days/week. All patients will be educated by physiotherapist to perform the movements for wrist, hand and arm in complete autonomy.In Control Group, these activates will be performed without any device.
  Interventions: Other: Usual care

INTERVENTIONS:
Device: Gloreha Aria — Device offers specific programs that help patients to move arm, wrist and fingers
  Arms: Treatment Group
Other: Usual care — Conventional occupational therapy
  Arms: Participants Usual Care (PUC)

SUMMARY:
Stroke is one of the leading causes of death and disability and has been described as a worldwide epidemic (1). Stroke survivors are affected by impairments and limitations of cognitive, language, perceptual, sensory, and motor functions. After a stroke, patients can improve spontaneously within the first 3 months (2) and then more slowly in the following year. The first day, decreased oedema and partial reperfusion of the ischemic penumbra may possibly explain these phenomena, but the improvement of neurological deficit in the following weeks suggests plasticity phenomena and brain cortical reorganization (3). While most recovery is thought to be made in the first few weeks after stroke, patients may make improvements on functional tasks many months after having a stroke (4). Restoring arm and hand skill after a stroke remains challenging, even though stroke rehabilitation programs have proven partial efficacy Repetitive task training has been shown to be effective in some aspects of rehabilitation, such as improving walking distance and speed and improving upper limb function (5).

In this project, the investigators will use "Gloreha ARIA" (7) a new sensor-based therapy device designed for motor recovery of impaired upper limb Gloreha Aria offers specific programs that help patients to move arm, wrist and fingers. Therapists can customize therapy by focusing on a specific motor task.

DETAILED DESCRIPTION:
The hypothesis was that rehabilitation with this device could be not inferior in comparison with hands-on physiotherapy, in the reeducation of upper arm in the patient affected by stroke from cerebral ischemia or hemorrhage that had occurred ≤ 30 days before.

The principle purpose of this study will be to evaluate:

1. The feasibility of this new device
2. Efficacy in improving arm function abilities in the rehabilitation of patients with stroke in the sub-acute phase.

Post-stroke patients admitted for inpatient rehabilitation to the Neurological Rehabilitation will be screened for enrolment and randomized in a controlled trial.

All the patients will be informed about the aim and experimental procedures before enrolment, thus written informed consent will be obtained from all of them. Patients included in the study will be randomly assigned to intervention or control group according to simple randomization technique (computerized random numbers).

ELIGIBILITY:
Inclusion Criteria:

* to exhibit first cerebral vascular disease with unilateral hemispherical lesion confirmed by CT scan or MRI;
* to be sub-acute patients (less than 30 days from the cerebral vascular event);
* being affected by upper limb paresis;

Exclusion Criteria:

1. unable to understand verbal instruction or motor commands;
2. unilateral neglect;
3. apraxia;
4. significant visual impairment;
5. unstable medical condition;
6. significant orthopedic limitation to the shoulder, elbow; wrist and hand;
7. upper arm peripherical nerve lesion;
8. neuromuscular or neurodegenerative diseases;
9. spasticity > 3 in according to the Modifies Ashworth Scale (3);

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline of FMA-UE (Fugl-Meyer assessment upper extremity). | From date of randomization (T0) until the to the end of the study (T1) after an intervention lasting over a period of about 6 weeks, assessed after 30 rehabilitation sessions, lasting 30 min/ day each and performed 5 days/week.
  Assessment of sensorimotor function.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Vanoglio, PT, Principal Investigator — Istituti Clinici Scientifici Maugeri
Locations (1):
- Istituti Clinici Scientifici Maugeri IRCCS, Pavia, Italy

REFERENCES:
- [Background] Bennett DA, Krishnamurthi RV, Barker-Collo S, Forouzanfar MH, Naghavi M, Connor M, Lawes CM, Moran AE, Anderson LM, Roth GA, Mensah GA, Ezzati M, Murray CJ, Feigin VL; Global Burden of Diseases, Injuries, and Risk Factors 2010 Study Stroke Expert Group. The global burden of ischemic stroke: findings of the GBD 2010 study. Glob Heart. 2014 Mar;9(1):107-12. doi: 10.1016/j.gheart.2014.01.001. PMID 25432120
- [Background] Maulden SA, Gassaway J, Horn SD, Smout RJ, DeJong G. Timing of initiation of rehabilitation after stroke. Arch Phys Med Rehabil. 2005 Dec;86(12 Suppl 2):S34-S40. doi: 10.1016/j.apmr.2005.08.119. PMID 16373138
- [Background] Chen R, Cohen LG, Hallett M. Nervous system reorganization following injury. Neuroscience. 2002;111(4):761-73. doi: 10.1016/s0306-4522(02)00025-8. PMID 12031403
- [Background] Teasell RW, Murie Fernandez M, McIntyre A, Mehta S. Rethinking the continuum of stroke rehabilitation. Arch Phys Med Rehabil. 2014 Apr;95(4):595-6. doi: 10.1016/j.apmr.2013.11.014. Epub 2014 Feb 14. PMID 24529594
- [Background] French B, Thomas LH, Coupe J, McMahon NE, Connell L, Harrison J, Sutton CJ, Tishkovskaya S, Watkins CL. Repetitive task training for improving functional ability after stroke. Cochrane Database Syst Rev. 2016 Nov 14;11(11):CD006073. doi: 10.1002/14651858.CD006073.pub3. PMID 27841442